CLINICAL TRIAL: NCT06038682
Title: Monitoring Anticoagulation With Argatroban in Patients on Extracorporeal Membrane Oxygenation for Severe Lung Failure Using Anti-FIIa. Monitoring Anticoagulation With Unfractionated Heparin in Patients on Extracorporeal Membrane Oxygenation for Severe Lung Failure Using Anti-FXa.
Brief Title: Monitoring Anticoagulation in Patients on ECMO for Severe Lung Failure
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: FNO-KARIM-Argatroban
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: ARDS; COVID-19
Keywords: ECMO; ARDS (acute respiratory distress syndrome); anticoagulation; thrombotic complications; LMWH (low-molecular-weight heparin); Argatroban
MeSH Terms: conditions — COVID-19; Acute Lung Injury | interventions — argatroban; Heparin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be obtained from patients in course of the routine care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Argatroban anticoagulation: Study subjects in this group will receive Argatroban anticoagulation.
  Interventions: Drug: Argatroban Injection
- Heparin anticoagulation: Study subjects in this group will receive Heparin anticoagulation.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Argatroban Injection — Argatroban will be administered to the study subjects in this group in order to achieve anticoagulation.
  Groups: Argatroban anticoagulation
Drug: Heparin — Heparin will be administered to the study subjects in this group in order to achieve anticoagulation.
  Groups: Heparin anticoagulation

SUMMARY:
A monocentric observational study evaluates the accuracy of anticoagulation monitoring in critically ill patients on ECLS (extracorporeal life support) using new markers of the effect of direct thrombin inhibitors and also the accuracy of anticoagulation monitoring in patients on unfractionated heparin using anti-Xa. A more accurate setting of anticoagulation may lead to a reduction in the number of serious bleeding and thrombotic complications in these patients.

DETAILED DESCRIPTION:
Anticoagulation using a direct thrombin inhibitor, argatroban, is one of the modern options for anticoagulation in patients on VV (veno-venous) ECMO (extracorporeal membrane oxygenation) support, and in 2021 the ECMO center of the University Hospital Ostrava changed the standard anticoagulation using UHF (unfractionated heparin) to anticoagulation using Argatroban as a new standard of routine care. Argatroban shows more stable levels and has a short half-life, and a number of foreign ECMO centers have been using Argatroban for a long time also as basic anticoagulation in all ECMO patients.

To monitor the effect of direct thrombin inhibitors, it is possible to use monitoring of anti-FIIa activity, which directly assesses the effect of the anticoagulant on thrombin activity. Anticoagulation with Argatroban may reduce the risk of serious bleeding complications. Target values of aPTT (Activated Partial Thromboplastin Time) and anti-FIIa can be determined according to ELSO (Extracorporeal Life Support Organization) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COVID-19
* ARDS according to the Berlin definition
* Veno-venous (VV) ECMO
* Full coagulation with Argatroban or heparin to an anti-FIIa value of 0.4-1.5 or aPTT 50-60

Exclusion Criteria:

- age under 18 years

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients on VV (veno-venous) ECMO on anticoagulation with Argatroban or heparin.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of aPTT values with anti-IIa and Argatroban dose in patients on VV ECMO | up to 2 weeks
  Comparison of correlation of aPTT and anti-IIa with dynamics of D dimer, FDP (fibrin degradation product) and acute phase reactants of ferritin, CRP (C-reactive protein) Correlation of bleeding complications with aPTT, anti-IIa, platelets
Comparison of apt and anti-Xa values and heparin dose in patients on VV ECMO | up to 2 weeks
  Comparison of correlation of aPTT and anti-Xa with dynamics of D dimer, FDP and acute phase reactants of ferritin, CRP

SECONDARY OUTCOMES:
Frequency and severity of bleeding complications | up to 2 weeks
  Comparison of frequency and severity of bleeding complications in patients on anticoagulation with Argatroban and heparin
Frequency and severity of thrombotic complications | up to 2 weeks
  Comparison of frequency and severity of thrombotic complications in patients anticoagulated with Argatroban and heparin
Consumption of blood products (in ml) | up to 2 weeks
  The consumption of blood products (volume in ml) in patients on Argatroban and heparin

CONTACTS AND LOCATIONS:
Overall Officials: Filip Burša, MD, Ph.D., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

REFERENCES:
- [Background] Al-Samkari H, Gupta S, Leaf RK, Wang W, Rosovsky RP, Brenner SK, Hayek SS, Berlin H, Kapoor R, Shaefi S, Melamed ML, Sutherland A, Radbel J, Green A, Garibaldi BT, Srivastava A, Leonberg-Yoo A, Shehata AM, Flythe JE, Rashidi A, Goyal N, Chan L, Mathews KS, Hedayati SS, Dy R, Toth-Manikowski SM, Zhang J, Mallappallil M, Redfern RE, Bansal AD, Short SAP, Vangel MG, Admon AJ, Semler MW, Bauer KA, Hernan MA, Leaf DE; STOP-COVID Investigators. Thrombosis, Bleeding, and the Observational Effect of Early Therapeutic Anticoagulation on Survival in Critically Ill Patients With COVID-19. Ann Intern Med. 2021 May;174(5):622-632. doi: 10.7326/M20-6739. Epub 2021 Jan 26. PMID 33493012
- [Background] Kowalewski M, Fina D, Slomka A, Raffa GM, Martucci G, Lo Coco V, De Piero ME, Ranucci M, Suwalski P, Lorusso R. COVID-19 and ECMO: the interplay between coagulation and inflammation-a narrative review. Crit Care. 2020 May 8;24(1):205. doi: 10.1186/s13054-020-02925-3. PMID 32384917
- [Background] Godier A, Clausse D, Meslin S, Bazine M, Lang E, Huche F, Cholley B, Hamada SR. Major bleeding complications in critically ill patients with COVID-19 pneumonia. J Thromb Thrombolysis. 2021 Jul;52(1):18-21. doi: 10.1007/s11239-021-02403-9. Epub 2021 Mar 1. PMID 33646501
- [Background] Gils C, Vinholt PJ, Nybo M. Falsely prolonged activated partial thromboplastin time - a pre- and post-analytical issue. Biochem Med (Zagreb). 2019 Feb 15;29(1):011001. doi: 10.11613/BM.2019.011001. Epub 2018 Dec 15. PMID 30591818
- [Background] Seelhammer TG, Plack D, Lal A, Nabzdyk CGS. COVID-19 and ECMO: An Unhappy Marriage of Endothelial Dysfunction and Hemostatic Derangements. J Cardiothorac Vasc Anesth. 2020 Dec;34(12):3193-3196. doi: 10.1053/j.jvca.2020.09.132. Epub 2020 Oct 2. No abstract available. PMID 33228917
- [Background] Alberio L, Angelillo-Scherrer A, Asmis L, Casini A, Fontana P, Graf L, Hegemann I, Kremer Hovinga JA, Korte W, Lecompte T, Martinez M, Nagler M, Studt JD, Tsakiris DA, Wuillemin W. Recommendations on the use of anticoagulants for the treatment of patients with heparin-induced thrombocytopenia in Switzerland. Swiss Med Wkly. 2020 Apr 24;150:w20210. doi: 10.4414/smw.2020.20210. eCollection 2020 Apr 20. PMID 32329806
- [Derived] Bursa F, Frelich M, Sklienka P, Nemcova S, Kucerova Z, Jor O, Romanova T, Konde A, Janosek J, Sagan J, Maca J. Activated Partial Thromboplastin Time and Anti-IIa Monitoring in Argatroban Anticoagulation in COVID-19 Patients on Venovenous Extracorporeal Membrane Oxygenation. Clin Appl Thromb Hemost. 2025 Jan-Dec;31:10760296251341315. doi: 10.1177/10760296251341315. Epub 2025 May 21. PMID 40396972